CLINICAL TRIAL: NCT02775214
Title: Conventional Direct Laryngoscopy Vs. Video Laryngoscopy With The C-MAC For Pyloromyotomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in staffing structure, no longer fit original study design
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Nicole Horn, pediatric anesthesiologist, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1306011553
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Results first posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Pyloric Stenosis; Intubation, Pediatric
Keywords: Storz C-MAC; direct laryngoscopy; pyloromyotomy; rapid sequence
MeSH Terms: conditions — Pyloric Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Direct Laryngoscopy (No Intervention): Endotracheal intubation will be performed by conventional direct laryngoscopy.
- Video Laryngoscopy (Active Comparator): Endotracheal intubation will be performed by video laryngoscopy with the C-MAC.
  Interventions: Device: Video Laryngoscopy

INTERVENTIONS:
Device: Video Laryngoscopy
  Other Names: C-MAC
  Arms: Video Laryngoscopy

SUMMARY:
The purpose of this study is to compare two different ways of placing breathing tubes for surgery. Both ways are used currently to place breathing tubes and are safe and effective. This study seeks to determine if one way is better than the other for infants with pyloric stenosis.

DETAILED DESCRIPTION:
Specific aims of this study include determining if there is a difference in the desaturation rates of the two different intubation techniques- Direct Laryngoscopy and the C-MAC video laryngoscope. Also is there a difference in intubation success between the two techniques, does intubation success vary with different training levels, and does desaturation rate differ among training levels.

ELIGIBILITY:
Inclusion Criteria:

* Need general anesthesia for pyloromyotomy procedure
* Have been informed of the nature of the study and informed consent has been obtained from the legally responsible guardian

Exclusion Criteria:

* Abnormal/difficult airway
* Allergy to succinylcholine and/or propofol

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2013-09; Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Horn, MD, Principal Investigator — Sponsor-Investigator
Locations (1):
- Riley Hospital for Children at IU Health, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4/19/17-7/12/22 pediatric hospital infants <6m with pyloric stenosis
Groups:
- Video Laryngoscopy: Endotracheal intubation will be performed by video laryngoscopy with the C-MAC.
  Video Laryngoscopy
Period: Overall Study
Arm/Group | Conventional Direct Laryngoscopy | Video Laryngoscopy
Started | 30 | 32
Completed | 28 | 32
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: <6m of age with pyloric stenosis
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Direct Laryngoscopy | Video Laryngoscopy | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 32 | 62
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex/Gender were not collected from any participant.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Pyloric Stenosis [Count of Participants; unit: Participants] | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Desaturation Below 80% During Intubation
Description: Patient had a desaturation below 80% during intubation with either conventional laryngoscope or video laryngoscope
Time Frame: During intubation attempt (less than two minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Direct Laryngoscopy | Video Laryngoscopy
Number analyzed (Participants) | 30 | 32
Participants | 6 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data was collected per patient from intubation through recovery period, a time frame of 24 hours
Description: Adverse event was defined as desaturation below 80% during intubation
Arm/Group | Conventional Direct Laryngoscopy | Video Laryngoscopy
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 6/30 | 4/32
Other Adverse Events (participants affected / at risk) | 0/30 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Direct Laryngoscopy (N=30) | Video Laryngoscopy (N=32)
desaturation (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) — desaturation below 80% during intubation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT02775214/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT02775214/ICF_001.pdf